CLINICAL TRIAL: NCT01834287
Title: Promoting Physical Activity in Latinas Via Interactive Web-Based Technology
Brief Title: Pasos Hacia La Salud - Physical Activity Intervention for Latinas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Dr.Bess Marcus, Professor and Chair, Department of Family and Preventive Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pasos Hacia La Salud; R01CA159954-02 (NIH)
Record Dates: First submitted 2013-04-12; First posted 2013-04-17 (Estimated); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Inactivity
Keywords: Physical Activity; Latinas; Web-based; Spanish-language
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physical Activity Intervention (Experimental): Motivationally-tailored, Spanish Language, Internet-based Physical Activity intervention that specifically addresses the Physical Activity barriers and intervention needs/preferences of Latinas.
  Interventions: Behavioral: Physical Activity Intervention
- Wellness Control (Active Comparator): Internet-based, Spanish language, Wellness Contact control intervention addressing relevant health topics other than Physical Activity.
  Interventions: Behavioral: Wellness Control

INTERVENTIONS:
Behavioral: Physical Activity Intervention — Participants in the Physical Activity intervention arm of the study receive a Spanish language, motivationally-tailored, Internet-based Physical Activity intervention that specifically addresses the Physical Activity barriers and intervention needs/preferences of Latinas.
  Arms: Physical Activity Intervention
Behavioral: Wellness Control — Participants will receive a Spanish language, Internet-based Wellness Contact control intervention addressing relevant health topics other than physical activity.
  Arms: Wellness Control

SUMMARY:
In this study, investigators are specifically targeting Latina women as they are more likely to be inactive and, therefore, are at higher risk for developing chronic conditions such as obesity, diabetes, or cardiovascular disease.

The objective of Pasos Hacia La Salud is to test a Spanish-language Internet-based Physical Activity Intervention, in comparison to a Spanish-language Internet-based Wellness Contact Control condition. Participants are randomly assigned to one of two groups (Exercise and General Wellness).

The investigators hypothesize that at the end of treatment, intervention participants will report significantly more minutes of moderate intensity physical activity per week than the wellness contact control participants.

DETAILED DESCRIPTION:
In the U.S., Latino women (Latinas) report higher rates of inactivity than their non-Hispanic White and male counterparts and thus are disproportionately burdened by related health conditions (e.g., cancer, hypertension, heart disease, stroke, diabetes). Cultural factors, socioeconomic circumstances, language and educational barriers limit Latinas access to public health interventions that promote physically active lifestyles. To address this public health crisis, effective interventions that leverage state-of-the-art theory and methods are needed to reach this at-risk population. Our research group has over 20 years experience developing and evaluating individually-tailored, computer expert system-driven, physical activity interventions (based on Social Cognitive Theory and the Transtheoretical Model) through various channels and settings. In our recent pilot (R21NR009864), we culturally and linguistically adapted our tailored intervention for sedentary Latinas and conducted a small randomized trial of the modified program (N=93). A total of 81 participants completed the 6-month study (87% retention) and increased their physical activity from a mean of 17 minutes per week (SD=25.76) at baseline to 147 minutes (SD=241.55) at six months whereas contact control participants increased their physical activity from 12 minutes per week (SD=21.99) at baseline to 97 minutes (SD=118.49) at six months. These observed improvements in physical activity in our intervention group, along with high retention rates, participant-reported desire for an Internet-delivered program, and formative work developing our program in an Internet format lend support for testing an Internet intervention tailored to the needs of Latinas. Therefore, for the current proposal, we will build on our previous work by conducting an adequately powered (N=200) randomized controlled trial to test the efficacy of our culturally and linguistically modified, individually tailored physical activity intervention delivered via the Internet relative to an Internet wellness contact control condition (including cardiovascular health information developed for Latinos by the NHLBI). Data will be collected at baseline, 6 months (post-treatment), and 12 months (maintenance) using well-established physical activity measures (7-Day PAR, Actigraphs), as well as a comprehensive set of psychosocial questionnaires. We hypothesize that at end of treatment (month six) intervention participants will report significantly more minutes of moderate intensity physical activity per week than the wellness contact control participants. We will also examine the maintenance of treatment effects at 12 months, potential mediators and moderators of the intervention-physical activity relationship, and the costs of delivering the tailored Internet program. In the proposed study we seek to promote physical activity among an underserved population using a high-reach, low-cost, technology-based strategy, which has great potential for adoption on a larger scale and thus high potential for reducing health disparities in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Generally healthy (If asthma and/or high blood pressure, may be able to participate with physician consent)
* Sedentary (Less than 60 minutes per week of moderate or vigorous physical activity)
* Latina (self-identified)
* Must be able to read and write Spanish fluently
* 18 - 65 years of age
* Planning on living in the area for the next 12 months
* Daily access to a computer with high speed internet

Exclusion Criteria:

* Pregnant or planning on becoming pregnant
* BMI greater than 45
* Not able to walk continuously for 30 minutes/limited ability to complete daily activity or ability to exercise
* Exercise is against advice of doctor
* Heart disease/treatment
* Heart murmur
* Angina/chest pain or Angina/chest pain with exertion
* Palpitations
* Stroke/Transient Ischemic Attacks
* Peripheral Vascular Disease
* Diabetes I or II
* Chronic Infectious Disease - HIV, Hepatitis
* Chronic liver disease
* Cystic Fibrosis
* Abnormal EKG on last EKG performed
* Emphysema, Chronic bronchitis, Chronic Obstructive Pulmonary Disease
* Seizure in past year
* Surgery in past year on heart, lung, joint, orthopedic surgery
* Surgery pending in next year on lung, joint, orthopedic surgery
* Unusual/concerning shortness of breath
* Asthma (may be able to participate with physician consent)
* High blood pressure/high blood pressure medication (may be able to participate with physician consent)
* Use of beta blockers
* Abnormal Medical Stress Test
* Musculoskeletal problems
* Fainting/dizziness more than 3 times in past year OR interferes with daily activities OR causes loss of balance
* Cancer treatment in past 3 months
* Hospitalized for psychiatric disorder in past 3 years or suicidal

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2011-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bess H Marcus, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California San Diego, La Jolla, California, United States

REFERENCES:
- [Derived] Larsen B, Dunsiger SI, Pekmezi D, Linke S, Hartman SJ, Marcus BH. Psychosocial mediators of physical activity change in a web-based intervention for Latinas. Health Psychol. 2021 Jan;40(1):21-29. doi: 10.1037/hea0001041. Epub 2020 Nov 23. PMID 33370154
- [Derived] Hartman SJ, Pekmezi D, Dunsiger SI, Marcus BH. Physical Activity Intervention Effects on Sedentary Time in Spanish-Speaking Latinas. J Phys Act Health. 2020 Mar 1;17(3):343-348. doi: 10.1123/jpah.2019-0112. PMID 32035412
- [Derived] Linke SE, Dunsiger SI, Gans KM, Hartman SJ, Pekmezi D, Larsen BA, Mendoza-Vasconez AS, Marcus BH. Association Between Physical Activity Intervention Website Use and Physical Activity Levels Among Spanish-Speaking Latinas: Randomized Controlled Trial. J Med Internet Res. 2019 Jul 24;21(7):e13063. doi: 10.2196/13063. PMID 31342902
- [Derived] Marquez B, Norman GJ, Fowler JH, Gans KM, Marcus BH. Weight and weight control behaviors of Latinas and their social ties. Health Psychol. 2018 Apr;37(4):318-325. doi: 10.1037/hea0000597. Epub 2018 Feb 1. PMID 29389157
- [Derived] Larsen B, Marcus B, Pekmezi D, Hartman S, Gilmer T. A Web-Based Physical Activity Intervention for Spanish-Speaking Latinas: A Costs and Cost-Effectiveness Analysis. J Med Internet Res. 2017 Feb 22;19(2):e43. doi: 10.2196/jmir.6257. PMID 28228368
- [Derived] Marcus BH, Hartman SJ, Larsen BA, Pekmezi D, Dunsiger SI, Linke S, Marquez B, Gans KM, Bock BC, Mendoza-Vasconez AS, Noble ML, Rojas C. Pasos Hacia La Salud: a randomized controlled trial of an internet-delivered physical activity intervention for Latinas. Int J Behav Nutr Phys Act. 2016 May 28;13:62. doi: 10.1186/s12966-016-0385-7. PMID 27234302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Physical Activity Intervention | Wellness Control
Started | 104 | 101
Completed | 90 | 94
Not Completed | 14 | 7

BASELINE CHARACTERISTICS:
Population: 205 eligible participants (13 ineligible post-randomization were removed from analysis)
Groups:
- Total: Total of all reporting groups
Arm/Group | Physical Activity Intervention | Wellness Control | Total
Number analyzed (Participants) | 104 | 101 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] — Age, years
  years | 38.84 (10.61) | 39.57 (10.36) | 39.20 (10.47)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex assigned at birth
  Participants
    Female | 104 | 101 | 205
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Self-reported Ethnicity
  Participants
    Hispanic or Latino | 104 | 101 | 205
    Not Hispanic or Latino | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Weekly Minutes of Physical Activity as Measured by the 7-Day PAR (Physical Activity Recall), From Baseline to 6-months and 12-months.
Description: The 7-Day PAR is an interviewer administered instrument that uses multiple strategies for increasing accuracy of participant recall regarding many types of activities such as time spent sleeping and moderate, hard, and very hard intensity activities. The 7-Day PAR is used across many studies assessing physical activity and has consistently demonstrated acceptable reliability, internal consistency, and congruent validity with other objective measures of activity levels.
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: minutes/week
Arm/Group | Physical Activity Intervention | Wellness Control
Number analyzed (Participants) | 104 | 101
minutes/week
  Baseline | 8.01 (14.95) | 10.44 (23.98)
  6 months | 112.83 (97.05) | 63.04 (88.33)
  12 months | 107.29 (106.46) | 74.64 (89.24)
Statistical Analysis 1: Comparison: Physical Activity Intervention vs Wellness Control; Test type: Superiority; p = .001, Regression, Linear; Mean Difference (Final Values) = 31.0, 95% CI 2-sided [9.6 to 52.4]

ADVERSE EVENTS:
Time Frame: baseline through 12m
Arm/Group | Physical Activity Intervention | Wellness Control
All-Cause Mortality (participants affected / at risk) | 0/104 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/104 | 0/101
Other Adverse Events (participants affected / at risk) | 0/104 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes